CLINICAL TRIAL: NCT03875950
Title: Standardized Patient Encounters to Improve Counseling for Pre-Exposure Prophylaxis (PrEP) for HIV Prevention to Adolescent Girls and Young Women (AGYW) in Kenya
Brief Title: Standardized Patient Encounters to Improve PrEP Counseling for Adolescent Girls and Young Women in Kenya
Acronym: PrIYA-SP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Pamela Kohler, Associate Professor, School of Nursing: Department Of Psychosocial And Community Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00005595; R01HD094630 (NIH)
Record Dates: First submitted 2019-02-15; First posted 2019-03-15 (Actual); Results first posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: HIV/AIDS
Keywords: Adolescents; Young women; HIV care and treatment; Clinical training; Africa; Kenya
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training intervention (Experimental): In this cluster randomized control trial design, the experimental arm refers to the 12 study sites that are randomly assigned to receive the clinician training intervention. The intervention is a clinician training using standardized patient actors to improve communication and empathy skills of health care workers who deliver PrEP to adolescent girls and young women to prevent HIV.
  Interventions: Behavioral: Clinician training intervention
- Standard of care control (No Intervention): In this randomized cluster randomized control trial design, the no intervention arm refers to the 12 study sites that are randomly assigned not to receive the clinician training intervention. Instead, these study sites will receive the standard of care, which is no standardized patient actor training, for health care workers who deliver PrEP to adolescent girls and young women to prevent HIV.

INTERVENTIONS:
Behavioral: Clinician training intervention — This intervention is a clinician training using standardized patient actors to improve communication and empathy skills of health care workers delivering PrEP to adolescent girls and young women to prevent HIV in Kenya.
  Arms: Training intervention

SUMMARY:
The goal of this study is to facilitate uptake of and adherence to HIV pre-exposure prophylaxis (PrEP) among adolescent girls and young women (AGYW) in Kenya. The investigators will conduct a cluster randomized controlled trial at 24 health facilities in Kisumu, Kenya of a clinical training intervention using standardized patient actors. The hypothesis is that the training will improve quality of PrEP service delivery, defined as adherence to national guidelines and non-judgmental communication.

DETAILED DESCRIPTION:
Despite global gains in female-controlled HIV prevention strategies, the incidence of HIV in adolescent girls and young women (AGYW) continues to rise. Pre-exposure prophylaxis (PrEP) has been shown to reduce the risk of HIV acquisition in trial settings, however real-world effectiveness at scale is limited by poor adherence.

An important barrier to uptake and adherence to HIV prevention services among AGYW is the experience of judgmental, and non-empathetic interactions with health care workers (HCWs). New strategies are needed to improve provider counseling and communication skills to support PrEP adherence among AGYW. Standardized patient actors (SPs) have been used in a variety of settings to improve clinical assessment and care skills, as well as patient outcomes.

The "PrIYA-SP" study aims to improve HCW communication skills and adherence to PrEP guidelines through a cluster randomized trial of a SP actor training intervention. Twenty-four facilities that currently offer PrEP to AGYW in Kisumu County, Kenya will be selected. The first phase will include a cross-sectional assessment by unannounced SPs who will present to clinics portraying AGYW seeking PrEP, according to case scripts. Following the baseline assessment, 12 facilities will be randomized to the SP training intervention. The two-day intervention consists of didactic sessions covering national guidelines and communication skills, values clarification exercises, role playing sessions with SPs, and a group debriefing with HCW participants. Following the intervention, unannounced SPs will repeat the cross-sectional assessment.

The primary outcome is quality of counseling, defined as adherence to national guidelines for PrEP delivery and use of non-judgmental communication skills. An intention-to-treat (ITT) analysis will be used to evaluate whether the SP training intervention resulted in higher quality counseling at intervention compared to control facilities, adjusted for relevant baseline characteristics and quality measures. The investigators hypothesize that this SP training intervention will improve quality delivery of PrEP to AGYW compared to standard of care.

Results from this study will directly inform operational guidelines for PrEP delivery to AGYW in low-resource settings and offer a potentially scalable strategy to improve PrEP service delivery and adherence among AGYW.

ELIGIBILITY:
Inclusion Criteria: Listed by population

Facilities:

* Facilities located in a county in Western Kenya
* Currently offering PrEP services to adolescent girls and young women

Health care workers:

* Age 18 or older
* Current employee of one of the 24 study sites
* Able to provide consent

Exclusion Criteria: Listed by population

Facilities:

* Health facilities where PrEP services are staffed by contract workers, program, or study staff

Health care workers:

* Study staff seconded to the site as part of a trial or intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2019-03-02 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela K Kohler, RN, MPH, PhD, Principal Investigator — University of Washington
Locations (1):
- Kenyatta National Hospital, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: Yes
The study investigators are prepared to share data with other researchers in accordance with NIH policies and other local regulations.
Supporting Information: Study Protocol
Time Frame: Summary data may be shared or otherwise made available to interested parties starting 6 months after publication of trial results
Access Criteria: Access to data will be determined on a case-by-base basis in agreement with the Kenyan Ministry of Health. De-identified data will be made available for secondary analyses. Any data sharing will be performed through secure servers and/or encrypted external drives.

REFERENCES:
- [Derived] Larsen A, Wilson KS, Kinuthia J, John-Stewart G, Richardson BA, Pintye J, Abuna F, Lagat H, Owens T, Kohler P. Standardised patient encounters to improve quality of counselling for pre-exposure prophylaxis (PrEP) in adolescent girls and young women (AGYW) in Kenya: study protocol of a cluster randomised controlled trial. BMJ Open. 2020 Jun 21;10(6):e035689. doi: 10.1136/bmjopen-2019-035689. PMID 32565464

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 232 providers consented to unannounced patient actor visits (125 at invention sites and 107 at control sites). The number of providers at intervention sites is higher than the number of providers trained, because all newly hired staff at health facilities provided consent during the outcome assessments which took place after the training.
Period: Overall Study
Arm/Group | Training Intervention | Standard of Care Control
Started | 125 | 107
Completed | 125 | 107
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Health providers of pre-exposure prophylaxis services at health facilities in Kenya
Groups:
- Total: Total of all reporting groups
Arm/Group | Training Intervention | Standard of Care Control | Total
Number analyzed (Participants) | 125 | 107 | 232
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 31 [28 to 36] | 31 [28 to 35] | 31 [28 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 59 | 134
  Male | 50 | 48 | 98
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 125 | 107 | 232
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Kenya | 125 | 107 | 232
Number of years providing HIV prevention services [Median (Inter-Quartile Range); unit: years] | 4 [2 to 7] | 3 [2 to 6] | 4 [2 to 6]
Prior receipt of HIV prevention training [Count of Participants; unit: Participants] | 54 | 52 | 106

OUTCOME MEASURES:

1. Primary Outcome: Quality of PrEP Counseling Provided by Health Care Workers Delivering PrEP to Adolescent Girls and Young Women for HIV Prevention in Kenya
Description: Quality is assessed as total score from a checklist provided by the SPs after each unannounced visit (n=71 SP visits in each arm) including domains of communication skills and adherence to national guidelines. Communication quality is assessed in an adapted version of the Bayer-Fetzer Kalamazoo Consensus Statement; scores range from 7-28 with higher scores indicating higher quality communication. Guideline adherence is assessed in a scoring system adapted from the Kenyan National AIDS & STI Control Programme guidelines; scores range from 0-13 with higher scores indicating higher PrEP competency. Each measure is computed as a percent of total score possible. The total quality score will be a combined continuous score and rescaled out of 100 per unannounced SP visit. Mean scores among all SP encounters taking place in facilities randomized to the clinical intervention will be compared to mean scores among those randomized to standard of care.
Time Frame: Unannounced standardized patient actor visits take approximately 15 minutes each, taking place over 3-4 months.
Population: Outcomes were assessed by unannounced patient actors who portrayed patients seeking PrEP services. There were 71 patient actor visits at control, and 71 patient actor visits at intervention sites. Visits were not matched to specific providers and some providers may have been seen twice, so the total number of providers evaluated is unknown.
Measure: Mean (Standard Deviation); unit: percentage of total score possible
Units Other Than Participants: USP visits
Groups:
- Training Intervention: In this cluster randomized control trial design, the experimental arm refers to the 12 study sites that are randomly assigned to receive the clinician training intervention. The intervention is a clinician training using standardized patient actors to improve communication and empathy skills of health care workers who deliver PrEP to adolescent girls and young women to prevent HIV.
  Clinician training intervention: This intervention is a clinician training using standardized patient actors to improve communication and empathy skills of health care workers delivering PrEP to adolescent girls and young women to prevent HIV in Kenya.
  Outcome measures are assessed through 71 unannounced patient actor visits.
- Standard of Care Control: In this randomized cluster randomized control trial design, the no intervention arm refers to the 12 study sites that are randomly assigned not to receive the clinician training intervention. Instead, these study sites will receive the standard of care, which is no standardized patient actor training, for health care workers who deliver PrEP to adolescent girls and young women to prevent HIV.
  Outcome measures are assessed through 71 unannounced patient actor visits.
Arm/Group | Training Intervention | Standard of Care Control
Number analyzed (Participants) | NA | NA
Number analyzed (USP visits) | 71 | 71
percentage of total score possible
  Overall quality | 73.6 (16.3) | 58.4 (16.7)
  Guideline adherence | 57.2 (25.4) | 36.2 (26.9)
  Communication skills | 90.0 (10.9) | 80.5 (11.4)

2. Secondary Outcome: Competency Score Measuring Quality of PrEP Counseling Provided by Health Care Workers During Clinical Training Intervention [Among Intervention Arm Only]
Description: The secondary outcome is PrEP competency among HCWs in interactions with SPs during the clinical training intervention, assessed as sub-scores for interpersonal skills, communication quality, and guideline adherence. Interpersonal skills are assessed using the Interpersonal skills (IPS) assessment tool (Van Zanten 2007); scores range from 1-16 with higher scores indicating better interpersonal skills. Communication quality is assessed in an adapted version of the Bayer-Fetzer Kalamazoo Consensus Statement; scores range from 7-28 with higher scores indicating higher quality communication. Guideline adherence is assessed in a scoring system adapted from the Kenyan National AIDS & STI Control Programme guidelines; scores range from 0-13 with higher scores indicating higher competency. The total competency score will be a combined continuous score (range 8-57) per SP interaction during the clinical training intervention. All scores are rescaled as a percent of total points possible.
Time Frame: Standardized patient actor training interactions take approximately 15 minutes each and will occur during a two-day training intervention. Trainings will be conducted over a period of 2-3 months.
Population: The 94 health providers who participated in the training intervention
Measure: Mean (Standard Deviation); unit: percentage of total score possible
Arm/Group | Training Intervention
Number analyzed (Participants) | 94
percentage of total score possible
  Overall quality (sum of adherence and communication) | 83.1 (10.1)
  Guideline adherence | 66.1 (20.7)
  Communication skills | 96.2 (8.1)
  Interpersonal skills | 86.9 (8.7)

ADVERSE EVENTS:
Time Frame: 18 months from initiation of the training intervention
Arm/Group | Training Intervention | Standard of Care Control
All-Cause Mortality (participants affected / at risk) | 0/125 | 0/107
Serious Adverse Events (participants affected / at risk) | 0/125 | 0/107
Other Adverse Events (participants affected / at risk) | 0/125 | 0/107

LIMITATIONS AND CAVEATS:
Intervention roll-out was delayed during the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-05-16): https://cdn.clinicaltrials.gov/large-docs/50/NCT03875950/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-08): https://cdn.clinicaltrials.gov/large-docs/50/NCT03875950/SAP_001.pdf